CLINICAL TRIAL: NCT05699850
Title: ARTIFICIAL INTELLIGENCE APPLICATIONS IN REPRODUCTIVE MEDICINE
Brief Title: ARTIFICIAL INTELLIGENCE IN REPRODUCTIVE MEDICINE
Acronym: AI in ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al Baraka Fertility Hospital (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, MD, consultant Doctor, Al-Azhar University
Other Study IDs: Kamal-AI
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: ARTIFICIAL INTELLIGENCE (AI) APPLICATIONS IN REPRODUCTIVE MEDICINE
Keywords: ARTIFICIAL INTELLIGENCE (AI); IVF; ART
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ARTIFICIAL INTELLIGENCE (AI) — ARTIFICIAL INTELLIGENCE (AI) APPLICATIONS IN REPRODUCTIVE MEDICINE

SUMMARY:
Many studies have been published investigating the use of AI as an unbiased, automated approach to embryo assessment. This review will summarize the recent AI advancements in the IVF field. Hopefully, that incorporating AI technology into the IVF clinics may be the next frontier in the journey towards personalised reproductive medicine and improved fertility outcomes for patients.

DETAILED DESCRIPTION:
ARTIFICIAL INTELLIGENCE (AI) APPLICATIONS IN REPRODUCTIVE MEDICINE

Kamaleldin Abdullah Rageh, M.D. (1).

Mohammad Atef Behery, M.D. (2)

Elsayed Ali Farag, M.D. (1)

1 -Department of Obstetrics and Gynecology, Faculty of medicine, Al-Azhar University, Cairo, Egypt.

2-International Islamic Center for Population Studies and Research, Al-Azhar University, Cairo, Egypt.

Abstract:

In spite of improved almost all aspects of IVF: ovarian stimulation, embryo culture and transfer, the pregnancy rates still not satisfactory. Studies confirm that up to 50% of the performed IVF cycles fail and there may be no direct explanation for this.

And it's worthy to mention that accurately predicting the outcome of an IVF cycle has yet to be achieved. One reason for this is the method of selecting an embryo for transfer. Morphological assessment of embryos is the traditional method of evaluating embryo quality and selecting which embryo to transfer. However, this subjective method of assessing embryos leads to inter- and intra-observer variability, resulting in less than optimal IVF success rates. Although time-lapse incubators and preimplantation genetic testing for aneuploidy have been introduced to help increase the chances of live birth, the outcomes remain less than ideal.

Currently, infertility treatments exert a lot of financial and emotional stress, especially in patients with previously failed IVF treatments, where there is no clear cause to be identified is a common, heartbreaking endpoint when the emotional, financial and physical burden of the treatment escalate to continue finding answers, but AI systems might help solve the dilemma by picking the best viable embryos that humans can't do. AI technologies have excellent potential to help the infertility field to soar over its current narrow focus on individual embryos and detect new patterns hidden in the patient data for overcoming the prevailing infertility cases.

The embryo selection is the most critical factor for the success of IVF. However, there is no single definitive criterion that can predict the success of an embryo. Rather, embryo selection is based on a variety of factors, making it is difficult to predict the probability of a successful pregnancy for each patient and to fully understand the cause of each failure. So, Utilization of artificial intelligence (AI) may support the clinicians in filling this knowledge gap, thereby being leveraged in the embryology laboratory to help improve IVF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* fertility related

Exclusion Criteria:

* fertile people

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: those people coming for fertility clinics
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
SUCCESS RATE | 4 MONTHS
  ARTIFICIAL INTELLIGENCE (AI) APPLICATIONS IN REPRODUCTIVE MEDICINE

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al-Azhar university, Cairo
  - Kamal Eldin Abdalla Rageh, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
will think about it